CLINICAL TRIAL: NCT01710033
Title: Phase 1, Placebo-controlled, Randomized, Sequential, Parallel-group, Dose Escalation Study to Evaluate 28-day Multiple Dose Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of CP-690,550 in Stable Renal Allograft Recipients
Brief Title: A Study Of CP-690,550 In Stable Kidney Transplant Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: A3921007
Record Dates: First submitted 2012-10-16; First posted 2012-10-18 (Estimated); Results first posted 2012-12-26 (Estimated); Last update posted 2012-12-26 (Estimated); Status verified 2012-11

CONDITIONS: Kidney Transplant
Keywords: CP-690,550; kidney transplant
MeSH Terms: interventions — tofacitinib; BID protein, human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- CP-690,550 5 mg BID (Experimental)
  Interventions: Drug: CP-690,550 5 mg BID
- CP-690,550 15 mg BID (Experimental)
  Interventions: Drug: CP-690,550 15 mg BID
- CP-690,550 30 mg BID (Experimental)
  Interventions: Drug: CP-690,550 30 mg BID

INTERVENTIONS:
Drug: Placebo — Placebo tables twice daily (BID) for 28 days
  Arms: Placebo
Drug: CP-690,550 5 mg BID — CP-690,550 5 mg BID for 28 days
  Arms: CP-690,550 5 mg BID
Drug: CP-690,550 15 mg BID — CP-690,550 15 mg BID for 28 days
  Arms: CP-690,550 15 mg BID
Drug: CP-690,550 30 mg BID — CP-690,550 30 mg BID for 28 days
  Arms: CP-690,550 30 mg BID

SUMMARY:
This was a Phase 1 dose escalation study to evaluate the safety, tolerability and pharmacokinetics of 28-day treatment of CP-690,550 in stable renal allograft recipients. In Stage 1, ascending doses of CP-690,550 were to be administered sequentially to 3-4 cohorts of subjects. After Stage 1, one dose level was to be selected for dosing in an expanded cohort in Stage 2.

ELIGIBILITY:
Inclusion Criteria:

* Medically stable kidney transplant patients 6 or more months after transplantation.
* Subjects must be on mycophenolate mofetil 1-2 gm daily
* In Cohort 3 (and 4, if conducted) in Stage 1 and the expanded cohort in Stage 2, subjects must be on a calcineurin inhibitor-free regimen.

Exclusion Criteria:

* Any rejection episodes in the preceding 3 months.
* Treated with Thymoglobulin or OKT3 for acute rejection in the past 6 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2003-09; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (8):
- United States (7):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Livingston, New Jersey
  - Pfizer Investigational Site, Madison, Wisconsin
- Pfizer Investigational Site

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921007&StudyName=A%20Study%20Of%20CP-690%2C550%20In%20Stable%20Kidney%20Transplant%20Patients

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo, Stage 1: Placebo matched to CP-690,550 tablet orally twice daily up to Day 28 followed by single oral dose on Day 29 in stable renal transplant recipients, receiving maintenance immunosuppression therapy (mycophenolate mofetil [MMF] with or without calcineurin inhibitor [cyclosporine {CsA} or tacrolimus {TAC}]) as per local clinical practice in Stage 1.
- CP-690,550 5 mg, Stage 1: CP-690,550 5 milligram (mg) tablet orally twice daily up to Day 28 followed by single oral dose on Day 29 in stable renal transplant recipients, receiving maintenance immunosuppression therapy (MMF), calcineurin inhibitor (CsA) as per local clinical practice in Stage 1.
- CP-690,550 15 mg, Stage 1: CP-690,550 15 mg tablet orally twice daily up to Day 28 followed by single oral dose on Day 29 in stable renal transplant recipients, receiving maintenance immunosuppression therapy (MMF), calcineurin inhibitor (CsA or TAC) as per local clinical practice in Stage 1.
- CP-690,550 30 mg, Stage 1: CP-690,550 30 mg tablet orally twice daily up to Day 28 followed by single oral dose on Day 29 in stable renal transplant recipients, receiving maintenance immunosuppression therapy (MMF) as per local clinical practice in Stage 1.
- CP-690,550 30 mg, Stage 2: CP-690,550 30 mg tablet orally twice daily up to Day 28 followed by single oral dose on Day 29 in stable renal transplant recipients, receiving maintenance immunosuppression therapy (MMF) as per local clinical practice in Stage 2.
Period: Stage 1
Arm/Group | Placebo, Stage 1 | CP-690,550 5 mg, Stage 1 | CP-690,550 15 mg, Stage 1 | CP-690,550 30 mg, Stage 1 | CP-690,550 30 mg, Stage 2
Started | 6 | 6 | 6 | 6 | 0
Completed | 6 | 6 | 6 | 6 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Stage 2
Arm/Group | Placebo, Stage 1 | CP-690,550 5 mg, Stage 1 | CP-690,550 15 mg, Stage 1 | CP-690,550 30 mg, Stage 1 | CP-690,550 30 mg, Stage 2
Started | 0 | 0 | 0 | 0 | 4
Completed | 0 | 0 | 0 | 0 | 3
Not Completed | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo, Stage 1: Placebo matched to CP-690,550 tablet orally twice daily up to Day 28 followed by single oral dose on Day 29 in stable renal transplant recipients, receiving maintenance immunosuppression therapy (MMF) with or without calcineurin inhibitor (CsA or TAC) as per local clinical practice in Stage 1.
- CP-690,550 30 mg, Stage 1 And 2: CP-690,550 30 mg tablet orally twice daily up to Day 28 followed by single oral dose on Day 29 in stable renal transplant recipients, receiving maintenance immunosuppression therapy (MMF) as per local clinical practice in Stage 1 and 2.
- Total: Total of all reporting groups
Arm/Group | Placebo, Stage 1 | CP-690,550 5 mg, Stage 1 | CP-690,550 15 mg, Stage 1 | CP-690,550 30 mg, Stage 1 And 2 | Total
Number analyzed (Participants) | 6 | 6 | 6 | 10 | 28
Age Continuous [Mean (Standard Deviation); unit: years] | 54.5 (15.0) | 53.0 (15.5) | 46.0 (17.8) | 54.2 (14.3) | 52.3 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3 | 2 | 8
  Male | 4 | 5 | 3 | 8 | 20

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) For CP-690,550
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast).
Time Frame: 0 (pre-dose), 0.5, 1, 2, 4, 8, 10, 12 hours post-dose on Day 1
Population: Analysis population included all randomized participants who received at least 1 dose of study treatment. Here "N" (Number of Participants Analyzed) signifies participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | CP-690,550 5 mg, Stage 1 | CP-690,550 15 mg, Stage 1 | CP-690,550 30 mg, Stage 1 And 2
Number analyzed (Participants) | 6 | 6 | 8
nanogram*hour per milliliter (ng*hr/mL) | 183 (75.3) | 754 (182) | 1200 (266)

2. Primary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) at Steady State For CP-690,550
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast) at steady state.
Time Frame: 0 (pre-dose), 0.5, 1, 2, 4, 8, 10, 12, 24 hours post-dose on Day 29
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | CP-690,550 5 mg, Stage 1 | CP-690,550 15 mg, Stage 1 | CP-690,550 30 mg, Stage 1 And 2
Number analyzed (Participants) | 6 | 6 | 9
ng*hr/mL | 319 (175) | 1300 (241) | 1560 (311)

3. Primary Outcome: Area Under the Curve From Time Zero to 12 Hour Concentration [AUC(0-12)] at Steady State For CP-690,550
Description: Area under the plasma concentration time-curve from zero to 12 hour concentration [AUC(0-12)] at steady state.
Time Frame: 0 (pre-dose), 0.5, 1, 2, 4, 8, 10, 12 hours post-dose on Day 29
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | CP-690,550 5 mg, Stage 1 | CP-690,550 15 mg, Stage 1 | CP-690,550 30 mg, Stage 1 And 2
Number analyzed (Participants) | 6 | 5 | 9
ng*hr/mL | 273 (132) | 1090 (150) | 1420 (253)

4. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) For CP-690,550
Time Frame: 0 (pre-dose), 0.5, 1, 2, 4, 8, 10, 12 hours post-dose on Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | CP-690,550 5 mg, Stage 1 | CP-690,550 15 mg, Stage 1 | CP-690,550 30 mg, Stage 1 And 2
Number analyzed (Participants) | 6 | 6 | 8
nanogram per milliliter (ng/mL) | 41.0 (14.9) | 140 (34.5) | 325 (113)

5. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) at Steady State For CP-690,550
Time Frame: 0 (pre-dose), 0.5, 1, 2, 4, 8, 10, 12, 24 hours post-dose on Day 29
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CP-690,550 5 mg, Stage 1 | CP-690,550 15 mg, Stage 1 | CP-690,550 30 mg, Stage 1 And 2
Number analyzed (Participants) | 6 | 5 | 9
ng/mL | 52.2 (15.2) | 220 (39.4) | 351 (46.3)

6. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) For CP-690,550
Time Frame: 0 (pre-dose), 0.5, 1, 2, 4, 8, 10, 12 hours post-dose on Day 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | CP-690,550 5 mg, Stage 1 | CP-690,550 15 mg, Stage 1 | CP-690,550 30 mg, Stage 1 And 2
Number analyzed (Participants) | 6 | 6 | 8
hours | 0.75 [0.50 to 2.00] | 1.50 [0.50 to 2.00] | 0.50 [0.50 to 2.00]

7. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) at Steady State For CP-690,550
Time Frame: 0 (pre-dose), 0.5, 1, 2, 4, 8, 10, 12, 24 hours post-dose on Day 29
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | CP-690,550 5 mg, Stage 1 | CP-690,550 15 mg, Stage 1 | CP-690,550 30 mg, Stage 1 And 2
Number analyzed (Participants) | 6 | 5 | 9
hours | 0.75 [0.50 to 2.00] | 0.50 [0.50 to 1.00] | 0.50 [0.50 to 1.00]

8. Primary Outcome: Accumulation Ratio (Rac) For CP-690,550
Description: Rac obtained from AUC(0-12) (Day 29) divided by AUC(0-12) (Day 1).
Time Frame: 0 (pre-dose), 0.5, 1, 2, 4, 8, 10, 12 hours post-dose on Day 1 and 29
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | CP-690,550 5 mg, Stage 1 | CP-690,550 15 mg, Stage 1 | CP-690,550 30 mg, Stage 1 And 2
Number analyzed (Participants) | 6 | 5 | 7
ratio | 1.48 (0.467) | 1.39 (0.245) | 1.22 (0.182)

9. Primary Outcome: Plasma Decay Half-Life (t1/2) For CP-690,550
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: 0 (pre-dose), 0.5, 1, 2, 4, 8, 10, 12 hours post-dose on Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | CP-690,550 5 mg, Stage 1 | CP-690,550 15 mg, Stage 1 | CP-690,550 30 mg, Stage 1 And 2
Number analyzed (Participants) | 4 | 2 | 8
hours | 3.36 (0.869) | NA (NA) — Data was not analyzed because there were not enough participants to perform a meaningful analysis. | 2.94 (0.620)

10. Primary Outcome: Plasma Decay Half-Life (t1/2) at Steady State For CP-690,550
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half at steady state.
Time Frame: 0 (pre-dose), 0.5, 1, 2, 4, 8, 10, 12, 24 hours post-dose on Day 29
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | CP-690,550 5 mg, Stage 1 | CP-690,550 15 mg, Stage 1 | CP-690,550 30 mg, Stage 1 And 2
Number analyzed (Participants) | 6 | 4 | 8
hours | 5.18 (2.00) | 5.15 (1.12) | 3.71 (0.201)

11. Primary Outcome: Mycophenolic Acid (MPA) Plasma Trough Concentration at Baseline
Description: Pro-drug MMF was metabolically converted to active form MPA in the liver. The baseline for MPA trough concentrations was defined as the average of the values obtained at Screening and on Day 1 (pre-dose). MPA levels were assessed at different visits to assess change in MPA trough levels due to CP-690,550 exposure.
Time Frame: Screening, 0 hour (pre-dose) on Day 1
Population: Analysis population included all randomized participants who received at least 1 dose of study treatment.
Measure: Mean (Standard Deviation); unit: Milligram per Liter (mg/L)
Arm/Group | Placebo, Stage 1 | CP-690,550 5 mg, Stage 1 | CP-690,550 15 mg, Stage 1 | CP-690,550 30 mg, Stage 1 And 2
Number analyzed (Participants) | 6 | 6 | 6 | 10
Milligram per Liter (mg/L) | 2.73 (1.23) | 2.18 (1.80) | 1.84 (1.13) | 2.43 (1.80)

12. Primary Outcome: Mycophenolic Acid (MPA) Plasma Trough Concentration at Day 8
Description: Pro-drug MMF was metabolically converted to active form MPA in the liver. MPA levels were assessed at different visits to assess change in MPA trough levels due to CP-690,550 exposure.
Time Frame: 0 hour (pre-dose) on Day 8
Population: Analysis population included all randomized participants who received at least 1 dose of study treatment.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Placebo, Stage 1 | CP-690,550 5 mg, Stage 1 | CP-690,550 15 mg, Stage 1 | CP-690,550 30 mg, Stage 1 And 2
Number analyzed (Participants) | 6 | 6 | 6 | 10
mg/L | 3.25 (2.77) | 2.11 (2.01) | 1.29 (0.48) | 2.56 (1.62)

13. Primary Outcome: Mycophenolic Acid (MPA) Plasma Trough Concentration at Day 15
Description: as for outcome 12
Time Frame: 0 hour (pre-dose) on Day 15
Population: Analysis population included all randomized participants who received at least 1 dose of study treatment.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Placebo, Stage 1 | CP-690,550 5 mg, Stage 1 | CP-690,550 15 mg, Stage 1 | CP-690,550 30 mg, Stage 1 And 2
Number analyzed (Participants) | 6 | 6 | 6 | 10
mg/L | 3.15 (1.75) | 2.36 (2.21) | 1.48 (0.63) | 2.74 (1.52)

14. Primary Outcome: Mycophenolic Acid (MPA) Plasma Trough Concentration at Day 29
Description: as for outcome 12
Time Frame: 0 hour (pre-dose) on Day 29
Population: Analysis population included all randomized participants who received at least 1 dose of study treatment.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Placebo, Stage 1 | CP-690,550 5 mg, Stage 1 | CP-690,550 15 mg, Stage 1 | CP-690,550 30 mg, Stage 1 And 2
Number analyzed (Participants) | 6 | 6 | 6 | 10
mg/L | 2.61 (1.77) | 2.68 (2.00) | 4.30 (3.88) | 3.24 (1.71)

15. Primary Outcome: Mycophenolic Acid (MPA) Plasma Trough Concentration at Day 57
Description: as for outcome 12
Time Frame: 0 hour (pre-dose) on Day 57
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Placebo, Stage 1 | CP-690,550 5 mg, Stage 1 | CP-690,550 15 mg, Stage 1 | CP-690,550 30 mg, Stage 1 And 2
Number analyzed (Participants) | 6 | 5 | 6 | 10
mg/L | 2.60 (1.56) | 2.89 (2.75) | 1.75 (1.10) | 2.67 (1.87)

16. Primary Outcome: Cyclosporine (CsA) Plasma Trough Concentration at Baseline
Description: The baseline for CsA trough concentrations was defined as the average of the values obtained at Screening and on Day 1 (pre-dose). CsA levels were assessed at different visits to assess change in CsA trough levels due to CP-690,550 exposure.
Time Frame: Screening, 0 hour (pre-dose) on Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo, Stage 1 | CP-690,550 5 mg, Stage 1 | CP-690,550 15 mg, Stage 1
Number analyzed (Participants) | 1 | 5 | 3
ng/mL | 249.50 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 81.00 (41.99) | 173.00 (51.11)

17. Primary Outcome: Cyclosporine (CsA) Plasma Trough Concentration at Day 8
Description: CsA levels were assessed at different visits to assess change in CsA trough levels due to CP-690,550 exposure.
Time Frame: 0 hour (pre-dose) on Day 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo, Stage 1 | CP-690,550 5 mg, Stage 1 | CP-690,550 15 mg, Stage 1
Number analyzed (Participants) | 1 | 4 | 3
ng/mL | 137.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 77.25 (47.28) | 134.00 (17.78)

18. Primary Outcome: Cyclosporine (CsA) Plasma Trough Concentration at Day 15
Description: CsA levels were assessed at different visits to assess change in CsA trough levels due to CP-690,550 exposure.
Time Frame: 0 hour (pre-dose) on Day 15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo, Stage 1 | CP-690,550 5 mg, Stage 1 | CP-690,550 15 mg, Stage 1
Number analyzed (Participants) | 1 | 5 | 3
ng/mL | 207.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 86.60 (43.71) | 160.33 (24.58)

19. Primary Outcome: Cyclosporine (CsA) Plasma Trough Concentration at Day 29
Description: CsA levels were assessed at different visits to assess change in CsA trough levels due to CP-690,550 exposure.
Time Frame: 0 hour (pre-dose) on Day 29
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo, Stage 1 | CP-690,550 5 mg, Stage 1 | CP-690,550 15 mg, Stage 1
Number analyzed (Participants) | 1 | 5 | 3
ng/mL | 226.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 96.00 (53.43) | 125.00 (22.34)

20. Primary Outcome: Cyclosporine (CsA) Plasma Trough Concentration at Day 57
Description: CsA levels were assessed at different visits to assess change in CsA trough levels due to CP-690,550 exposure.
Time Frame: 0 hour (pre-dose) on Day 57
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo, Stage 1 | CP-690,550 5 mg, Stage 1 | CP-690,550 15 mg, Stage 1
Number analyzed (Participants) | 1 | 5 | 3
ng/mL | 292.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 91.20 (72.71) | 152.00 (43.28)

21. Primary Outcome: Tacrolimus (TAC) Plasma Trough Concentration at Baseline
Description: The baseline for TAC trough concentrations was defined as the average of the values obtained at Screening and on Day 1 (pre-dose). TAC levels were assessed at different visits to assess change in TAC trough levels due to CP-690,550 exposure.
Time Frame: Screening, 0 hour (pre-dose) on Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo, Stage 1 | CP-690,550 15 mg, Stage 1
Number analyzed (Participants) | 2 | 3
ng/mL | 6.75 (2.47) | 7.17 (1.76)

22. Primary Outcome: Tacrolimus (TAC) Plasma Trough Concentration at Day 8
Description: TAC levels were assessed at different visits to assess change in TAC trough levels due to CP-690,550 exposure.
Time Frame: 0 hour (pre-dose) on Day 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo, Stage 1 | CP-690,550 15 mg, Stage 1
Number analyzed (Participants) | 2 | 3
ng/mL | 7.50 (2.12) | 8.00 (1.00)

23. Primary Outcome: Tacrolimus (TAC) Plasma Trough Concentration at Day 15
Description: TAC levels were assessed at different visits to assess change in TAC trough levels due to CP-690,550 exposure.
Time Frame: 0 hour (pre-dose) on Day 15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo, Stage 1 | CP-690,550 15 mg, Stage 1
Number analyzed (Participants) | 2 | 3
ng/mL | 8.00 (2.83) | 6.67 (2.08)

24. Primary Outcome: Tacrolimus (TAC) Plasma Trough Concentration at Day 29
Description: TAC levels were assessed at different visits to assess change in TAC trough levels due to CP-690,550 exposure.
Time Frame: 0 hour (pre-dose) on Day 29
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo, Stage 1 | CP-690,550 15 mg, Stage 1
Number analyzed (Participants) | 2 | 3
ng/mL | 7.00 (2.83) | 12.67 (4.51)

25. Primary Outcome: Tacrolimus (TAC) Plasma Trough Concentration at Day 57
Description: TAC levels were assessed at different visits to assess change in TAC trough levels due to CP-690,550 exposure.
Time Frame: 0 hour (pre-dose) on Day 57
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo, Stage 1 | CP-690,550 15 mg, Stage 1
Number analyzed (Participants) | 2 | 3
ng/mL | 5.00 (1.41) | 6.33 (0.58)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Placebo, Stage 1 | CP-690,550 5 mg, Stage 1 | CP-690,550 15 mg, Stage 1 | CP-690,550 30 mg, Stage 1 And 2
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/6 | 2/6 | 1/10
Other Adverse Events (participants affected / at risk) | 5/6 | 5/6 | 5/6 | 8/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo, Stage 1 (N=6) | CP-690,550 5 mg, Stage 1 (N=6) | CP-690,550 15 mg, Stage 1 (N=6) | CP-690,550 30 mg, Stage 1 And 2 (N=10)
Gastroenteritis (Infections and infestations) | 0 | 0 | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo, Stage 1 (N=6) | CP-690,550 5 mg, Stage 1 (N=6) | CP-690,550 15 mg, Stage 1 (N=6) | CP-690,550 30 mg, Stage 1 And 2 (N=10)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 2
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gingival hyperplasia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Catheter site haemorrhage (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 2 | 0 | 0
Cytomegalovirus viraemia (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 1 | 2
Laryngitis (Infections and infestations) | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0 | 0
Onychomycosis (Infections and infestations) | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 1 | 0 | 0
Tinea versicolour (Infections and infestations) | 0 | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 1 | 0
Reticulocyte count decreased (Investigations) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 3 | 0 | 1
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.